CLINICAL TRIAL: NCT05368818
Title: An Analysis of the Improvement and Quality of Life Trends for UK/ROI Patients Treated With Cosentyx (Secukinumab) in a Retrospective Analysis of the BADBIR Data Source
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457AGB06
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Plaque Psoriasis
Keywords: Cosentyx,; Secukinumab,; Quality of Life,; UK
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- All patients: Included all patients prescribed an on-label secukinumab dose
  Interventions: Other: Secukinumab
- Patients with Psoriatic Arthritis (PsA): Included patients classified as having a concomitant PsA diagnosis, if it was declared in the Baseline table
  Interventions: Other: Secukinumab

INTERVENTIONS:
Other: Secukinumab — Included patients treated with Cosentyx (Secukinumab) in a retrospective analysis of the BADBIR data source
  Other Names: Cosentyx

SUMMARY:
This was a retrospective, observational study of psoriasis patients treated with secukinumab, using secondary data from BADBIR. BADBIR is a UK/ROI pharmacovigilance registry that was initiated in 2007 to monitor the long-term safety of biologic drugs used to treat psoriasis. The study used longitudinal data within the registry to track the trends relating to the disease. For the analysis of improvement and patient reported QoL, patients with a minimum of one follow-up visit were included. The index date was defined as the date of initiation of secukinumab treatment, and follow-up visits were at 6-, 12-, 18-, & 24-months post-index.

DETAILED DESCRIPTION:
The BADBIR data was current up until the 31st August 2019 for this analysis.

Study period: From 1st July 2015, as secukinumab was included in BADBIR in January 2016 and patients backdated 6 months, to 31st August 2019.

Identification period: From 1st July 2015 to 31st August 2019 was used to identify applicable patients for analysis.

Index date: Initiation of secukinumab treatment within the BADBIR database.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the biologic cohort:

* Age ≥18 years at initiation of secukinumab.
* At least one follow-up visit post-registry enrollment.
* On-label dosing of secukinumab of 300mg.

Inclusion criteria for the PsA biologic cohort:

* Age ≥18 years at initiation of secukinumab.
* At least one follow-up visit post-registry enrollment.
* On-label dosing of secukinumab of 300mg.
* Diagnosis of PsA at baseline.

Exclusion Criteria:

- The patient did not meet the criteria stated above.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The BADBIR registry included patients treated for psoriasis using biologics, conventional systemic therapies, or small molecule immunomodulators
Sampling Method: Non-Probability Sample
Enrollment: 767 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reporting high/very high QoL changes from Baseline (BL) (from 2 or 3 at BL to 0) | throughout the study, approximately 4 years (1st July 2015 to 31st August 2019 )
  Patient reported QoL for five specific DLQI domains from baseline up to 24 months of UK/ROI psoriasis patients enrolled in BADBIR who were initiated on secukinumab treatment were reported.
  Following 5 domains were included:
  * Embarrassment and/or self conciousness
  * Social leisure
  * Work/study
  * Problems relating to partner, friends and relatives
  * Sexual difficulties

SECONDARY OUTCOMES:
Age | Baseline
  Age was reported
Sex | Baseline
  Sex information was reported
Ethinicity | Baseline
  Ethinicity information was reported
Employment status | Baseline
  Employment status was reported
Smoking Characteristics | Baseline
  Smoking characteristics were reported
Weight | Baseline
  Weight information was reported
Height | Baseline
  Height information was reported
Body Mass Index (BMI) | Baseline
  BMI information was reported
Waist circumference | Baseline
  Waist information was reported
Absolute Psoriasis Area Severity Index (aPASI) at BL | Baseline
  aPASI scores were reported
Total Dermatology Life Quality Index (DLQI) at BL | Baseline
  Total DLQI score was reported
DQLI Domain - 2) embarrassment and/or self-consciousness - proportion of those who reported high or very high at baseline | Baseline
  DQLI Domain - 2) embarrassment and/or self-consciousness - proportion of those who reported high or very high at baseline were reported
DQLI Domain - 5) social and leisure activities - proportion of those who reported high or very high at baseline | Baseline
  DQLI Domain - 5) social and leisure activities - proportion of those who reported high or very high at baseline were reported
DQLI Domain - 7) work/study - proportion of those who reported high or very high at baseline | Baseline
  DQLI Domain - 7) work/study - proportion of those who reported high or very high at baseline were reported
DQLI Domain - 8) problems relating to partner, friends, and relatives - proportion of those who reported high or very high at baseline | Baseline
  DQLI Domain - 8) problems relating to partner, friends, and relatives - proportion of those who reported high or very high at baseline were reported
DQLI Domain - 9) sexual difficulties - proportion of those who reported high or very high at baseline | Baseline
  DQLI Domain - 9) sexual difficulties - proportion of those who reported high or very high at baseline were reported
Number of Biologic naïve/experienced patients | Baseline
  Patients were listed as being previously experienced to a biologic treatment if a drug name listed in 'Biologics_Drugname', was listed as a 'DrugName' in the DrugPastTherapy table. If a patient had no record of a biologic drugname in the DrugPastTherapy table, the patient was recorded as biologic naive.
Number of Psoriatic Arthritis (PsA) patients | Baseline
  Patients were classified as Psoriatic Arthritis using the 'PsoriaticArthritis' flag in the Baseline_Psoriasis tables. (0=No, 1=Yes, Null=not entered).
Time to PsA diagnosis | Baseline
  Time to PsA onset was calculated using the 'PsoriaticArthritisOnset' variable from the FupPsoriasis table and 'YearOnset' from the Baseline Psoriasis table. The time to PsA diagnosis was reported as the difference between 'PsoriaticArthritisOnset' minus 'YearOnset'.
Number of patients with No PsA and nail involvement | Baseline
  Patients were classified as having nail involvement using the 'NailsNumber' variable from the Baseline_Psoriasis table
Number of nails involved | Baseline
  Number of nails involved were reported
Number of patients with at least one Comorbidity | Baseline
  Comorbidities were derived from the MedDRA Preferred Term (PT) variable in the BaselineComorbidities table. If a patient recorded at least one comorbidity, listed within the available data, this patient was recorded as "Has a comorbidity".
Number of patients with five most common comorbidities at BL | Baseline
  Comorbidities were derived from the MedDRA Preferred Term (PT) variable in the BaselineComorbidities table. If a patient recorded at least one comorbidity, listed within the available data, this patient was recorded as "Has a comorbidity". The top 5 comorbidities at baseline were determined via highest frequency of occurrence by cohort and were reported for each subgroup
Frequency of on-label 300mg prescription | Baseline
  Frequency of on-label 300mg prescription was categorized into the following, N/A (new convention for licensed dose), Once a week (induction), Once monthly & Once every four weeks. To determine if the patients were on-label, confirmation was required that the right dosage was being given; patients were included as on-label if they reported a dose value of 300 using the 'Dose' and the unit mg with the 'DoseUnit' variable in the DrugBiologicTherapy table. The frequency of prescription was assessed using the 'Frequency' variable and mapped in accordance with the following categories: N/A (new convention for licensed dose), Once a week (induction), Once monthly, once every four weeks or Not reported.
Proportion of PsA subjects with a total DLQI score of >10 | throughout the study, approximately 4 years (1st July 2015 to 31st August 2019)
  Proportion of PsA subjects with a total DLQI score of >10 at baseline achieving a score of 0 or 1 at 6-month intervals to 24 months (window of +/- 60 days), stratified by none, any, <5 nails, ≥5 nails or all nails involved at baseline was reported.
Proportion of PsA patients with an aPASI score of 0, <=1, <=2 or <=3 | throughout the study, approximately 4 years (1st July 2015 to 31st August 2019)
  Proportion of PsA patients with an aPASI score of 0, <=1, <=2 or <=3 at each 6-month interval up to 24 months (window of +/-60 days), stratified by none, any, <5 nails, ≥5 nails or all nails involved at baseline was reported.
Proportion of Psoriasis patients with an aPASI score of 0, <=1, <=2 or <=3 | throughout the study, approximately 4 years (1st July 2015 to 31st August 2019)
  Proportion of Psoriasis patients with an aPASI score of 0, <=1, <=2 or <=3 at each 6-month interval up to 24 months (window of +/-60 days), stratified by patients being biologic naive or biologic experienced was reported.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CAIN457AGB06 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17932